CLINICAL TRIAL: NCT01528670
Title: Monitoring of Patients Treated With Particle Therapy Using Positron-Emission-Tomography (PET): The MIRANDA Study.
Acronym: MIRANDA
Status: Withdrawn | Type: Observational
Why Stopped: Administrative barriers
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Other Study IDs: MIRANDA
Record Dates: First submitted 2011-12-30; First posted 2012-02-08 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Particle Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Skull Base
- Lower GI
- Prostate
- Pelvic Region
- Head-and-Neck
- Upper GI
- Brain
- Other

SUMMARY:
The purpose of this clinical study is to investigate the clinical feasibility and effectiveness of off-line Positron-Emission-Tomography (PET) quality assurance for promoting the accuracy of proton and carbon ion beam therapy. One main clinical advantage of ion therapy over conventional radiation therapy is the excellent conformation of the delivered dose to the tumour volume while well sparing the surrounding healthy tissue. However, clinical exploitation of this potential to the maximum extent requires in-vivo validation of the actual treatment delivery and, in particular, of the ion beam range within the patient. Since the primary ions are completely stopped in the target volume as opposed to photon radiation, no conventional quality assurance techniques like transmission electronic portal imaging can be applied to monitor ion beam therapy. Hence, ion treatment planning currently relies on models and experimental data accurately validated in tissue-equivalent targets, but no direct verification of the actual treatment delivery and of the ion beam range within the patient is possible in standard clinical practice.

At present, PET offers the unique possibility to monitor the precision of ion irradiation in-vivo and non-invasively. The method is based on the detection of the b+-activity which is formed as a by-product of the irradiation, i.e. without administration of radio-tracers to the patient. A positive clinical impact of in-beam (i.e. during the irradiation) PET monitoring has been demonstrated for carbon ion therapy in the pilot project at GSI Darmstadt, Germany, and promising clinical data of post-radiation PET/CT imaging have been recently reported for passive proton beam delivery in USA and Japan. Therefore, a pilot clinical study is hereby proposed at the Heidelberg Ion Therapy Center in order to 1) assess the applicability of post-radiation PET imaging to scanned ion beam delivery, 2) identify the patient population which may benefit from it and 3) extract population-based information on the reliability of the beam range in different tumour locations for all the ion species clinically available at HIT.

The investigated patients are expected to benefit from this study, since in case of detected deviations between planned and actual treatment delivery a proper correction could be applied in the next irradiation fraction, assuring an overall better treatment than without any monitoring. Moreover, site-specific patient-population information on the ion range precision at HIT might enable improvement of the CT-range calibration curve as well as safe reduction of the treatment margins to promote enhanced treatment plan conformality for full clinical exploitation of the promises of ion beam therapy.

ELIGIBILITY:
Inclusion Criteria

* The patient is treated at the Heidelberger Ionenstrahl Therapiezentrum (HIT) with protons or carbon ions.
* During the radiotherapeutic treatment patient positioning is verified using validated radiological imaging such as cone beam CT, X-ray or conventional CT (Reference-Imaging as described above).
* The patient is at least 18 years of age and is able to give informed consent.
* The patient has been informed about the aims and the content of the study.

Exclusion Criteria

* No informed consent to take part in the study.
* Medical reasons that impair the patients from being in the supine position for the data acquisition time, e.g. pain.
* Non-compliance of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Particle Therapy at the Heidelberg Ion Therapy (HIT) Center will be included and grouped into 8 anatomical regions: Brain, Skull base, Head-and-neck, Upper GI, Lower GI, Prostate, Pelvic region and other.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
TBA | TBA
  TBA

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E Combs, MD, Principal Investigator — University Hospital of Heidelberg
Locations (1):
- Department of Radiation Oncology, Heidelberg, Germany

REFERENCES:
- [Derived] Combs SE, Bauer J, Unholtz D, Kurz C, Welzel T, Habermehl D, Haberer T, Debus J, Parodi K. Monitoring of patients treated with particle therapy using positron-emission-tomography (PET): the MIRANDA study. BMC Cancer. 2012 Apr 3;12:133. doi: 10.1186/1471-2407-12-133. PMID 22471947